CLINICAL TRIAL: NCT01458444
Title: Acute Respiratory Failure After Cardio Thoracic Surgery: Non Invasive Ventilation (VNI) by BIPAP Vision Versus OPTIFLOW System, Comparison.
Brief Title: BIPAP Vision Versus OPTIFLOW System Comparison in Acute Respiratory Failure After Cardio Thoracic Surgery
Acronym: OPTIFLOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Collaborators: Hôpital NOVO (Other); Hopital Jean Minjoz (Other); University Hospital, Bordeaux (Other); University Hospital, Clermont-Ferrand (Other); Hopital Louis Pradel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SC11-007; 2011-A00125-36 (Other: ANSM)
Record Dates: First submitted 2011-10-21; First posted 2011-10-24 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Respiratory Insufficiency
Keywords: Respiratory Insufficiency; Cardiothoracic Surgery; Ventilation system
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BIPAP (Active Comparator): Non invasive ventilation (VNI) by BIPAP® vision
  Interventions: Device: Non invasive ventilation (VNI)
- OPTIFLOW (Experimental): OPTIFLOW system
  Interventions: Device: Non invasive ventilation

INTERVENTIONS:
Device: Non invasive ventilation (VNI) — BIPAP® vision
  Arms: BIPAP
Device: Non invasive ventilation — OPTIFLOW system
  Arms: OPTIFLOW

SUMMARY:
The OPTIFLOW ™ use is becoming more common in acute respiratory failure cases, but its place in relation to VNI (Bi-PAP mode) is not yet defined. OPTIFLOW ™ vs the VNI comparison of the use, in the immediate postoperative period, should lead to define the role of each technique and lead to a optimal rationalization of patients management with acute respiratory failure after surgery.

DETAILED DESCRIPTION:
Main objective: to determine, if the initiation of OPTIFLOW™ system immediate after cardio/ thoracic surgery with acute respiratory failure or immediate after post extubation in patients at risk, is not less than the start a VNI per BIPAP Vision ®system. In terms of reintubation rates, refusal to continue the technique, or switch to another technique proposed.

Secondary objectives:

* To assess changes in the sensation of dyspnea
* To analyze the skin tolerance and the comfort in this population
* To analyze the evolution of hemodynamic and respiratory parameters
* To compare the number of bronchoscopy performed during the patient's stay in intensive care unit
* Assess the number of postoperative pneumonia and antibiotic consumption
* To determine whether the initiation of any treatment changes in the immediate postoperative length of stay in intensive care and comprehensive.

ELIGIBILITY:
Inclusion Criteria:

* Patients after cardiac/thoracic surgery with acute respiratory failure defined by the presence of the following criteria:

  * report PaO2/FiO2 <300
  * Respiratory rate> 25 for at least 2 hours
  * Getting involved accessory respiratory muscles
  * paradoxical breathing Or
* In immediate after extubation, the patient will be eligible if present in the withdrawal test:

  * SaO2 <90% in 12 L of O2 during a trial of spontaneous ventilation tube on
  * PaO2 <10 kPa at a FiO2 ≥ 50% during a VS trial + pressure support
  * The presence of a risk factor: Obesity (BMI> 30), FEVG <40%, Failed extubation prior, stridor

Exclusion Criteria:

* Previous history of SAS
* Patient tracheotomy
* Comas non hypercapnic
* bradypnea
* Cardiac arrest
* Gastric Surgery recent
* Restlessness, lack of cooperation
* Nausea, vomiting
* Hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 830 (Actual)
Dates: Start 2011-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Failure of the ventilation system | One week
  Failure defined by reintubation rate, refusal to continue the technique, or switch to an another technique proposed breakdown

SECONDARY OUTCOMES:
Sensation of dyspnea | one week
Skin tolerance and comfort | One week
Evolution of hemodynamic and respiratory parameters | one week
number of bronchoscopy performed during the patient's stay in Intensive Care Unit | one week
number of postoperative pneumonia and antibiotic use | one week
length of stay in intensive care | one week

CONTACTS AND LOCATIONS:
Overall Officials: François STEPHAN, MD, Principal Investigator — CCML
Locations (1):
- Centre Chirurgical MarieLannelongue, Le Plessis-Robinson, Île-de-France Region, France

REFERENCES:
- [Derived] Stephan F, Barrucand B, Petit P, Rezaiguia-Delclaux S, Medard A, Delannoy B, Cosserant B, Flicoteaux G, Imbert A, Pilorge C, Berard L; BiPOP Study Group. High-Flow Nasal Oxygen vs Noninvasive Positive Airway Pressure in Hypoxemic Patients After Cardiothoracic Surgery: A Randomized Clinical Trial. JAMA. 2015 Jun 16;313(23):2331-9. doi: 10.1001/jama.2015.5213. PMID 25980660